CLINICAL TRIAL: NCT03679377
Title: Mandibular Slotplates
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Universitair Ziekenhuis Brussel (Other)
Responsible Party: Principal Investigator, Veerle Van Mossevelde, Director, Universitair Ziekenhuis Brussel
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: Mandi slot plates v 1.0
Record Dates: First submitted 2018-09-19; First posted 2018-09-20 (Actual); Last update posted 2019-08-28 (Actual); Status verified 2019-08

CONDITIONS: Craniofacial Abnormalities
Keywords: Orthognathic surgical procedures; Osteosynthesis
MeSH Terms: conditions — Craniofacial Abnormalities

STUDY DESIGN:
Intervention Model Description: Mandibular slotplates are placed during the osteosynthesis phase of the BSSO surgery. After clinical testing during the surgery the plates are removed and the osteotomy is fixated with bicortical screws.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Mandibular slotplate (Experimental): Mandibular slotplates are placed during BSSO surgery and their clinical usefullness is tested. Afterwards the plates are removed and the osteotomy is fixated by three bicortical screws.
  Interventions: Device: Mandibular slotplate

INTERVENTIONS:
Device: Mandibular slotplate — Mandibular slotplates are placed during the osteosynthesis phase of the BSSO surgery. After testing of the plates they are removed and the osteotomy is fixated with three bicortical screws.

SUMMARY:
A new osteosynthesis system for orthognathic surgery was proposed.This system allows small intra-operative adjustments of the bone fragments during the osteosynthesis phase of the operation (also known as the slot principle). Another possible advantage are the slant screw holes with chamfered ridges allowing easy placements of the screws via the small incision wound without undercuts in between the plate and the screwheads.

DETAILED DESCRIPTION:
Initial slotplates were developed for Le Fort I osteotomies, zygoma 'sandwich 'osteotomies and genioplasties. Those plates allowed for the slot principle to be performed during orthognathic surgery. Mandibular slotplates for bilateral sagittal split osteotomy (BSSO) were recently designed. The aim of the study is to evaluate their clinical usefulness and the applicability of the slot principle with these plates in BSSO.

ELIGIBILITY:
Inclusion Criteria:

• Patients undergoing single osteotomy BSSO surgery

Exclusion Criteria:

• Concomitant surgeries at the same time.

Ages: 12 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 9 (Estimated)
Dates: Start 2018-11-07 (Actual); Primary Completion 2019-12-31 (Estimated); Study Completion 2020-02-01 (Estimated)

PRIMARY OUTCOMES:
Feasebility of the slotprinciple | during surgery
  yes or no
Inclination of the screws | during surgery
  Useful yes or no

CONTACTS AND LOCATIONS:
Overall Officials: Brandaan Zigterman, MD, Principal Investigator — Universitair Ziekenhuis Brussel; Maurice Mommaerts, Prof Mult, Study Director — Universitair Ziekenhuis Brussel
Locations (1):
- universitair Ziekenhuis Brussel, Jette, Vlaams Brabant, Belgium